CLINICAL TRIAL: NCT04601012
Title: Optical Coherence Tomography Angiography in Patients Affected by SARS-CoV-2 Infection: a Pilot Study
Brief Title: OCTA Study: Retinal Vascular Changes in Patients With SARS-CoV-2 Infection
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gilda Cennamo, Principal Investigator, Federico II University
Other Study IDs: 2020/03
Record Dates: First submitted 2020-10-22; First posted 2020-10-23 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2020-10

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with COVID19: The patients with previous diagnosis of COVID19
  Interventions: Diagnostic Test: Optical coherence tomography angiography
- Control subjects: Healthy subjects without actual and previous ocular diseases
  Interventions: Diagnostic Test: Optical coherence tomography angiography

INTERVENTIONS:
Diagnostic Test: Optical coherence tomography angiography — Each subject underwent optical coherence tomography angiography to evaluate the retinal vessel density.

SUMMARY:
This study evaluates the retinal vascular features using optical coherence tomography angiography in patients that have been affected by COVID-19.

DETAILED DESCRIPTION:
To investigate the potential role of optical coherence tomography angiography in identifying the changes in retinal vessel density in patients that have been affected by COVID-19.

The optical coherence tomography angiography represents a noninvasive diagnostic technique that allows a detailed analysis of retinal vascular features.

ELIGIBILITY:
Inclusion Criteria:

* age older than 18 years
* diagnosis of previous COVID-19
* absence of previous ocular surgery, congenital eye disease, high myopia (>6 dioptres), actual or previous diagnosis of glaucoma, optic disc anomaly, macular or vitreoretinal diseases.
* absence of significant lens opacities, low-quality OCT and OCT-A images.

Exclusion Criteria:

* age younger than 18 years
* absence of previous diagnosis of COVID-19
* presence of previous ocular surgery, congenital eye disease, high myopia (>6 dioptres), actual or previous diagnosis of glaucoma, optic disc anomaly, macular or vitreoretinal diseases.
* presence of significant lens opacities, low-quality OCT and OCT-A images.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The participans were older than 18 years with previous diagnosis of COVID-19. They did not present other ophthalmological diseases.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-09-20 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-10-22 (Actual)

PRIMARY OUTCOMES:
The measurements of retinal features in patients with previous diagnosis of COVID19, using optical coherence tomography angiography. | one month
  The parameter analyzed by optical coherence tomography angiography was: retinal vessel density

CONTACTS AND LOCATIONS:
Overall Officials: Gilda Cennamo, Principal Investigator — Federico II University
Locations (1):
- University of Naples "Federico II", Naples, Italy